CLINICAL TRIAL: NCT04024644
Title: Third Molar: Evaluation of Caries, Periodontal Disease and Quality of Life and Its Variation Concerning to Dental Position
Brief Title: Third Molar: Caries, Periodontal Disease and Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Waldyr Antônio Jorge, PhD, clinical professor, University of Sao Paulo
Other Study IDs: Third molar Re
Record Dates: First submitted 2019-07-13; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Caries; Periodontal Diseases
Keywords: third molar; dental caries; periodontal disease; quality of life
MeSH Terms: conditions — Periodontal Diseases; Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Caries and periodontal disease are chronic diseases of the oral cavity. The incidence of caries and periodontal disease can vary depending on the position of the third molar, The aim of this study was to verify possible associations between oral health-related quality of life (QoL), periodontal disease, caries lesions and the position of the lower third molar.

DETAILED DESCRIPTION:
Caries and periodontal disease are chronic diseases of the oral cavity. The presence of third molar teeth can lead to periodontal disease in the region, and often can lead to injuries and damage to the oral health, having a significant impact on the quality of life. The incidence of caries and periodontal disease can vary depending on the position of the third molar. Purpose: The aim of this study was to verify possible associations between oral health-related quality of life (QoL), periodontal disease, caries lesions and the position of the lower third molar. Materials and Methods: The investigators performed a clinical, observational cross-sectional study within 116 patients that were screened attending to evaluate the need for extraction of third molars at of the specialization course of Oral and Maxillofacial Surgery of Dental School Foundation of University of São Paulo (FFO-USP). Caries, periodontal disease and quality of life are the outcomes that were evaluated by the main researcher. Caries lesions were assessed by visual tactile examination and periodontal disease through two probing sites around third molar, considering the presence of periodontal pathology when at least one periodontal probing depth was greater than 4 mm, and both were evaluated by radiograph diagnostic methods. The assessment of oral health related quality of life by Oral Health impact Profile questionary (OHIP-14), applied as an interview. The evaluation of the position of the third molars was made by clinical and panoramic radiographs according to the classification of Pell and Gregory and Winter. Data was treated and analyzed according to STATA 13.0, software with descriptive and inferential statistics. The level of significance used was 95%. The study had the approval of ethics committee from University of Sao Paulo Dental School (number 280084).

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiology (ASA) I patients (negative medical history)
* with at least one third molar erupted or partially erupted

Exclusion Criteria:

* systemically compromised
* allergic
* pregnants
* patients who had the four third molars included
* patients who have already undergone the extraction of one of the third molars

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants with at least one third molar erupted or partially erupted. , regardless of age, gender, cultural level or socioeconomic status could participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Caries | throughout study completion on average of one year
  Caries were assessed by visual tactile examination, only on occlusal surface in erupted or partially erupted third molars (visual tactile examination) and evaluation of the presence of the image on the panoramic radiograph.

SECONDARY OUTCOMES:
periodontal disease | throughout study completion on average of one year
  Periodontal disease was assessed by gingival sulcus probing in the third molars at two points: mesiobuccal and distobuccal regions. We considered the presence of Dp when the pocket was bigger than or equal to 4 mm.
Position of the lower third molars | throughout study completion on average of one year
  Position of the lower third molars were assessed by panoramic radiography, according to the classification of Pell and Gregory and Winter, performed by only one evaluator, following the criteria of imaginary lines as proposed by Almendros-Marques, et al.
Oral health related quality of life: Brazilian version of OHIP-14 questionnaire | throughout study completion on average of one year
  Oral health related quality of life (OHRQoL) were assessed by Brazilian version of OHIP-14 questionnaire. This instrument consists of 14 items arranged in 7 factors: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The answers were given corresponding to a total of 5 points on a Likert-type scale. The scale included the following responses: never (coded 0), hardly ever (coded 1), occasionally (coded 2), fairly often (coded 3), and very often (coded 4). The OHIP-14 scale ranged from 0 to 56, with higher scores indicating poorer QoL

CONTACTS AND LOCATIONS:
Overall Officials: Waldyr A. Jorge, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: 10.1016/j.joms.2011.09.034 — https://www.ncbi.nlm.nih.gov/pubmed/22177812
- Available data/document: Clinical Study Report: 10.1016/j.joms.2011.09.034 — https://www.ncbi.nlm.nih.gov/pubmed/31149009